CLINICAL TRIAL: NCT00713505
Title: A Behavioral Intervention Trial for Parents of Childhood Cancer Survivors With Neurobehavioral Late Effects
Brief Title: Educational and Skills Training Program for Parents of Childhood Cancer Survivors Who Have Neurobehavioral Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sunita Patel, City of Hope Medical Center
Allocation: Randomized
Other Study IDs: CDR0000598114; R03CA130731 (NIH); P30CA033572 (NIH); CHNMC-07250
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Cancer Survivor; Cognitive/Functional Effects; Leukemia; Long-term Effects Secondary to Cancer Therapy in Children; Lymphoma; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; long-term effects secondary to cancer therapy in children; cancer survivor; cognitive/functional effects; childhood acute lymphoblastic leukemia; childhood acute myeloid leukemia in remission; childhood anaplastic large cell lymphoma; childhood large cell lymphoma; childhood lymphoblastic lymphoma; childhood small noncleaved cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Lymphoma, Extranodal NK-T-Cell | interventions — Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (parent intervention program and usual care) (Experimental): Child participants and their families may access multidisciplinary psychosocial services (i.e., usual care). Parents also receive 8 weekly face-to-face training sessions (75-90 minutes each) with a therapist over approximately 2-3 months. Phone support/assistance is provided by the therapist within 2-3 days following each training session and then every 2 weeks for up to 6 months after completion of the training sessions.
  Interventions: Other: educational intervention; Procedure: psychosocial assessment and care
- Arm II (wait-list/usual care control [UCC]) (Active Comparator): Child participants and their families undergo usual care as in arm I and are placed on a wait-list.
  Interventions: Procedure: psychosocial assessment and care

INTERVENTIONS:
Other: educational intervention — Parents receive face-to-face training sessions with a therapist over approximately 2-3 months. Phone support/assistance is provided by the therapist within 2-3 days following each training session and then every 2 weeks for up to 6 months after completion of the training sessions.
  Arms: Arm I (parent intervention program and usual care)
Procedure: psychosocial assessment and care — Child participants and their families may access multidisciplinary psychosocial services (i.e., usual care).

SUMMARY:
RATIONALE: An educational and skills training program for the parent of a childhood cancer survivor with neurobehavioral dysfunction may help improve the child's school performance, thinking ability, and behavior.

PURPOSE: This randomized clinical trial is studying an educational and skills training program for parents of childhood cancer survivors who have neurobehavioral dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility of implementing an educational and skills training intervention for parents of a childhood cancer survivor with neurobehavioral dysfunction using face-to-face training sessions and phone assistance.
* To pilot test and collect preliminarily data on the indirect therapeutic impact of the parent training intervention on the child's academic, cognitive, and behavioral functioning.
* To pilot test and collect preliminary outcomes of the parent training intervention on parents of a childhood cancer survivor with neurobehavioral dysfunction.

OUTLINE: Parent and child participants are randomized to 1 of 2 intervention arms.

* Arm I (parent intervention program and usual care): In addition to medical care, child participants and their families may access multidisciplinary psychosocial services (i.e., usual care). Parents also receive 8 weekly face-to-face training sessions (75-90 minutes each) with a therapist over approximately 2-3 months. The training sessions include integration and didactic review of a parent's role as a behavioral and emotional support system for the child's school success; a parent's role as a monitor and motivator for school performance; a parent's role as an intervener and teacher of effective learning and study strategies; and a parent's role as a child advocate and accessor of educational and community resources. Parents are instructed to engage in ≥ 30 minutes of cognitive and academic activities with their child ≥ 4 days a week. The therapist will observe the parent (in the home or clinic) apply knowledge and techniques learned in the parent training sessions directly with the child at least once after the 4th parent-therapist session to provide feedback to the parent and child and to assess which parents may require more intense training and support. The sessions may be videotaped by the parent and provided to the therapist for review and follow up.

Phone support/assistance is provided by the therapist within 2-3 days following each training session to provide additional problem-solving assistance and teaching support to the parents while they are implementing the knowledge and strategies learned during the training sessions and to measure study adherence and behavioral implementation between the sessions. After completion of the training sessions, continued phone support/assistance is provided by the therapist every 2 weeks for up to 6 months to provide ongoing support and problem-solving and teaching assistance as needed and to promote ongoing maintenance of the trained parenting practices with a greater degree of independence. "Booster" in-person sessions may also occur if determined to be needed by both the therapist and parent.

* Arm II (wait-list/usual care control [UCC]): Child participants and their families undergo usual care as in arm I and are placed on a wait-list.

Parent and child participants in both arms complete battery testing and questionnaires at baseline, 3 months, and 6 months. Battery testing includes the Wechsler Individual Achievement Test (WIAT-II) and the WISC-IV Working Memory Index and Children's Memory Scale (CMS) subtests. Questionnaires include parent, teacher, and child [self-report] questionnaires (BASC-II, BRIEF, and SMALSI); Parent Behaviors Questionnaire-Revised; Parent Knowledge and Efficacy Questionnaire; and Parent's Treatment Barriers and Satisfaction Questionnaire.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Childhood cancer survivor who received CNS-directed therapy (i.e., intrathecal chemotherapy and/or cranial radiotherapy) for leukemia or non-Hodgkin lymphoma

  * In remission AND completed treatment ≥ 3 months ago
  * No brain tumors
* Enrolled in school and demonstrates a deficit (operationalized as at least one standard deviation below the age expected mean) on at least one objective test of attention or memory on baseline cognitive assessment screening AND has evidence of problems in learning and adaptive functioning

  * Parent, teacher, or self-report of problems as measured by a T-score of ≥ 60 on the BRIEF or BASC or below average academic achievement scores
  * Able to be tested in English using standardized cognitive and academic achievement tools

PATIENT CHARACTERISTICS:

* Primary participating parent or caregiver fluent in English and lives with the child
* No known history of a major psychiatric condition (i.e., psychosis) that precludes study participation (child or participating parent or caregiver)
* No history of child developmental disability prior to cancer diagnosis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
WIAT-II-Reading, Mathematics, and Writing composite scores as measured at baseline and 6 months (child participant)
Knowledge, efficacy, and self-report of pro-learning behaviors as measured by the PKEQ and PBQ-R at baseline, 3 months, and 6 months (parent participant)

SECONDARY OUTCOMES:
Parent, teacher, and self-report measures as measured by the BRIEF, BASC-II, and SMALSI at baseline, 3 months, and 6 months (child participant)
Performance on attention and memory tests as measured by the CMS and WISC-IV subtests at baseline and 6 months (child participant)
Parenting stress as measured by the PSI at baseline, 3 months, and 6 months (parent participant)

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Patel, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States